CLINICAL TRIAL: NCT03300050
Title: A Phase 1, Randomized, Controlled, Observer-blind Study to Assess the Reactogenicity, Safety, and Immunogenicity of a Live Attenuated Universal Influenza Vaccine (cH8/1N1 LAIV) Administered as a Single Priming Dose Followed Three Months Later by a Single Booster Dose of an Inactivated Universal Influenza Vaccine (cH5/1N1 IIV) (Adjuvanted With AS03A or Unadjuvanted) in 18 Through 39 Year-old Healthy Subjects, Contrasted With a Two Dose Schedule of an Inactivated Universal Influenza Vaccine (cH8/1N1 IIV + AS03A Followed Three Months Later by cH5/1N1 IIV + AS03A)
Brief Title: Safety and Immunogenicity of a Live-attenuated Universal Flu Vaccine Followed by an Inactivated Universal Flu Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Children's Hospital Medical Center, Cincinnati (Other); Duke University (Other); The Emmes Company, LLC (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVIA 057 (1082166-1)
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-07

CONDITIONS: Influenza; Vaccine
Keywords: live attenuated influenza vaccine; inactivated influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — AS03 adjuvant; Saline Solution

STUDY DESIGN:
Intervention Model Description: Eligible enrolled subjects will be randomized to any of the treatment arms (LAIV-IIV, Groups 1, 2, and 3; or IIV-IIV, Groups 4 and 5) under one allocation sequence, stratified by site, to allow comparability between study groups, such as LAIV-IIV vs IIV-IIV regimens (Groups 1 vs 4). Groups 1-3 will be inpatient and receive either LAIV or placebo as nasal drops at Dose 1. Groups 4-5 ill be outpatient and receive either IIV or placebo as an injection at Dose 1.
Who Masked: Participant, Care Provider, Investigator
Masking Description: An unblinded pharmacist will prepare Dose 1 and Dose 2. Participants and study staff will remain blinded to their exact treatment group but will be unblinded to their overall group allocation (inpatient or outpatient).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + adjuvant (Experimental): Participants received 0.5 mL cH8/1N1 LAIV administered as 0.25 mL drops per nostril on Day 1 followed by 0.5 mL AS03-adjuvanted cH5/1N1 IIV administered as an intramuscular injection on Day 85.
  Interventions: Biological: cH8/1N1 LAIV; Biological: AS03-adjuvanted cH5/1N1 IIV
- Group 2: cH8/1N1 LAIV and cH5/1N1 IIV (Experimental): Participants received 0.5 mL cH8/1N1 LAIV administered as 0.25 mL drops per nostril on Day 1 followed by 0.5 mL cH5/1N1 IIV administered as an intramuscular injection on Day 85.
  Interventions: Biological: cH8/1N1 LAIV; Biological: cH5/1N1 IIV
- Group 3: Placebo (Placebo Comparator): Participants received 0.5 mL of normal saline administered as 0.25 mL drops per nostril on Day 1 followed by 0.5 mL phosphate buffered saline (PBS) administered as an intramuscular injection on Day 85.
  Interventions: Biological: Normal saline; Biological: Phosphate buffered saline (PBS)
- Group 4: cH8/1N1 IIV + adjuvant and cH5/1N1 IIV + adjuvant (Experimental): Participants received 0.5 mL AS03-adjuvanted cH8/1N1 IIV administered as an intramuscular injection on Day 1 followed by 0.5 mL AS03-adjuvanted cH5/1N1 IIV administered as an intramuscular injection on Day 85.
  Interventions: Biological: AS03-adjuvanted cH5/1N1 IIV; Biological: AS03-adjuvanted cH8/1N1 IIV
- Group 5: Placebo (Placebo Comparator): Participants received 0.5 mL PBS administered as an intramuscular injection on Day 1 followed by 0.5 mL PBS administered as an intramuscular injection on Day 85.
  Interventions: Biological: Phosphate buffered saline (PBS)

INTERVENTIONS:
Biological: cH8/1N1 LAIV — Live-attenuated influenza virus vaccine (LAIV) expressing chimeric hemagglutinin (HA) with the H8 head and H1 stalk and neuraminidase (NA) subtype 1 (N1) (cH8/1N1):
  HA head, A/mallard/Sweden/24/2002 (H8N4); HA stalk, A/California/04/2009 (H1N1); NA, A/California/04/2009 (H1N1) containing the backbone of the cold-adapted/temperature sensitive of the Russian LAIV A/Leningrad/134/17/1957 (Len17 IDCDCRG46D).
  Administered intranasally as drops at a dose of 10⁷·⁵ (plus or minus ⁰·⁵) 50% egg infectious dose (EID50), formulated in a total volume of 0.5 mL sterile saline (0.25 mL per nostril).
  Arms: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + adjuvant; Group 2: cH8/1N1 LAIV and cH5/1N1 IIV
Biological: AS03-adjuvanted cH5/1N1 IIV — Chimeric H5 head with H1 stalk plus N1 (cH5/1N1) split virion inactivated influenza virus vaccine (IIV) plus AS03 adjuvant: HA head, A/Vietnam/1203/2004 (H5N1); HA stalk, A/California/04/2009 (H1N1); NA, A/California/04/2009 (H1N1).
  Administered intramuscularly at a dose of 15 μg of hemagglutinin in a volume of 0.5 mL of phosphate buffered saline (PBS).
  Other Names: cH5/1N1 IIV + AS03 adjuvant
  Arms: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + adjuvant; Group 4: cH8/1N1 IIV + adjuvant and cH5/1N1 IIV + adjuvant
Biological: cH5/1N1 IIV — Chimeric H5 head with H1 stalk plus N1 (cH5/1N1) split virion inactivated influenza virus vaccine (IIV):
  HA head, A/Vietnam/1203/2004 (H5N1); HA stalk, A/California/04/2009 (H1N1); NA, A/California/04/2009 (H1N1).
  Administered intramuscularly at a dose of 15 μg of hemagglutinin in a volume of 0.5 mL of phosphate buffered saline (PBS).
  Arms: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV
Biological: AS03-adjuvanted cH8/1N1 IIV — Chimeric H8 head with H1 stalk plus N1 (cH8/1N1) inactivated influenza vaccine plus AS03 adjuvant: HA head, A/mallard/Sweden/24/2002 (H8N4); HA stalk, A/California/04/2009 (H1N1); NA, A/California/04/2009 (H1N1).
  Administered intramuscularly at a dose of 15 μg of hemagglutinin in a volume of 0.5 mL of phosphate buffered saline (PBS).
  Other Names: cH8/1N1 IIV + AS03 adjuvant
  Arms: Group 4: cH8/1N1 IIV + adjuvant and cH5/1N1 IIV + adjuvant
Biological: Normal saline — Administered intranasally as 0.25 mL nasal drops per nostril
  Arms: Group 3: Placebo
Biological: Phosphate buffered saline (PBS) — Administered intramuscularly as 0.5 mL injection
  Arms: Group 3: Placebo; Group 5: Placebo

SUMMARY:
The clinical study will evaluate safety and the immune response of a prime- boost regimen with a live attenuated influenza vaccine (LAIV) prime and an inactivated split influenza vaccine (IIV) boost with or without adjuvant.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, controlled, observer-blind, Phase 1 trial in healthy male and female adults 18 through 39 years of age to evaluate safety and the immune response of a prime boost regimen with LAIV prime and IIV boost with or without adjuvant. Participants will be randomized 4:3:1:3:2 to one of five groups to receive a first dose of study cH8/1N1 LAIV (or placebo) or study cH8/1N1 IIV + AS03A adjuvant (or placebo) followed three months later by study cH5/1N1 IIV +/- AS03A adjuvant (or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand planned study procedures and demonstrate comprehension of the protocol procedures and knowledge of study by passing a written examination prior to vaccination.
* In the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* Male or non-pregnant female between, and including, 18 and 39 years of age at the time of the first vaccination.
* Healthy subjects without acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality*.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential must have a negative pregnancy test within 24 hours of vaccination.
* Female subjects of childbearing potential must have practiced adequate contraception for 30 days prior to first vaccination and agree to continue adequate contraception until 2 months after completion of the vaccination series (Month 5).
* Male subjects must be surgically sterile (e.g., vasectomy) or agree to practice adequate contraception from the first vaccination until 2 months after completion of the vaccination series (Month 5). Please refer to the glossary of terms for the definition of adequate contraception.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Medically diagnosed deviated nasal septum or nasal obstruction.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within 6 months before the first dose.
* Administration of long-acting immune-modifying drugs (e.g., infliximab, rituximab) within 6 months before the first dose (Visit 03), or planned administration any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose (Visit 03) up to Month 15 (Visit 15)
* Persons who should be annually vaccinated against influenza who live with or care for persons at high risk for influenza-related complications.
* History of influenza vaccination within 6 months prior to study enrollment or unwillingness to forego seasonal influenza vaccination during the entire study period.
* History of vaccination with an investigational pandemic influenza vaccine other than an 2009 H1N1 Pandemic (H1N1pdm09) vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Infection with human immunodeficiency virus regardless of clinical stage of immunodeficiency.
* History of current infection with hepatitis B virus or hepatitis C virus regardless of clinical presentation.
* History of or current autoimmune disease.
* Subjects diagnosed with excessive daytime sleepiness or narcolepsy; or history of narcolepsy in a subject's parent or sibling.
* History of Guillain-Barré syndrome.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines (including egg proteins); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Hypersensitivity to latex.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccines or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or male planning to father a child or either planning to discontinue contraceptive precautions.
* Current smoker.
* During screening, have a positive test for opiates without a prescription.
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
* Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
* Blood donation or planned blood donation within 30 days prior to the study vaccination through 30 days after the last blood drawn for this study.
* Have signs or symptoms that could confound or confuse assessment of study vaccine reactogenicity.
* Any hematological or biochemical parameter that is out of range of normal, and is considered clinically significant by the investigator.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bernstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Jeffrey Guptill, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meade P, Strohmeier S, Bermudez-Gonzalez MC, Garcia-Sastre A, Palese P, Simon V, Krammer F. Antigenic Landscape Analysis of Individuals Vaccinated with a Universal Influenza Virus Vaccine Candidate Reveals Induction of Cross-Subtype Immunity. J Virol. 2023 Jan 31;97(1):e0107022. doi: 10.1128/jvi.01070-22. Epub 2022 Dec 19. PMID 36533948
- [Derived] Nachbagauer R, Feser J, Naficy A, Bernstein DI, Guptill J, Walter EB, Berlanda-Scorza F, Stadlbauer D, Wilson PC, Aydillo T, Behzadi MA, Bhavsar D, Bliss C, Capuano C, Carreno JM, Chromikova V, Claeys C, Coughlan L, Freyn AW, Gast C, Javier A, Jiang K, Mariottini C, McMahon M, McNeal M, Solorzano A, Strohmeier S, Sun W, Van der Wielen M, Innis BL, Garcia-Sastre A, Palese P, Krammer F. A chimeric hemagglutinin-based universal influenza virus vaccine approach induces broad and long-lasting immunity in a randomized, placebo-controlled phase I trial. Nat Med. 2021 Jan;27(1):106-114. doi: 10.1038/s41591-020-1118-7. Epub 2020 Dec 7. PMID 33288923
- [Derived] Bernstein DI, Guptill J, Naficy A, Nachbagauer R, Berlanda-Scorza F, Feser J, Wilson PC, Solorzano A, Van der Wielen M, Walter EB, Albrecht RA, Buschle KN, Chen YQ, Claeys C, Dickey M, Dugan HL, Ermler ME, Freeman D, Gao M, Gast C, Guthmiller JJ, Hai R, Henry C, Lan LY, McNeal M, Palm AE, Shaw DG, Stamper CT, Sun W, Sutton V, Tepora ME, Wahid R, Wenzel H, Wohlbold TJ, Innis BL, Garcia-Sastre A, Palese P, Krammer F. Immunogenicity of chimeric haemagglutinin-based, universal influenza virus vaccine candidates: interim results of a randomised, placebo-controlled, phase 1 clinical trial. Lancet Infect Dis. 2020 Jan;20(1):80-91. doi: 10.1016/S1473-3099(19)30393-7. Epub 2019 Oct 17. PMID 31630990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community and enrolled at Cincinnati Children's Hospital Medical Center (Cincinnati, OH, USA) and the Duke Early Phase Clinical Research Unit (Durham, NC, USA) between October 10, 2017, and November 27, 2017.
Pre-assignment Details: Participants were randomly assigned in a 4:3:1:3:2 ratio to one of five treatment groups. Randomization was blocked (block size 13) and stratified by site. Participants received two sequential study vaccinations, an initial priming dose on Day 1 followed by a booster dose on Day 85.
Groups:
- Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant: Participants received 0.5 mL chimeric H8/1N1 live-attenuated influenza virus vaccine (cH8/1N1 LAIV) administered as 0.25 mL drops per nostril on Day 1 followed by 0.5 mL AS03 (Adjuvant System 03)-adjuvanted chimeric H5/1N1 inactivated influenza virus vaccine (cH5/1N1 IIV) administered as an intramuscular injection on Day 85.
- Group 3: Placebo: Participants received 0.5 mL normal saline administered as 0.25 mL drops per nostril on Day 1 followed by 0.5 mL phosphate buffered saline (PBS) administered as an intramuscular injection on Day 85.
- Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant: Participants received 0.5 mL AS03-adjuvanted chimeric H8/1N1 inactivated influenza vaccine (cH8/1N1 IIV) administered as an intramuscular injection on Day 1 followed by 0.5 mL AS03-adjuvanted cH5/1N1 IIV administered as an intramuscular injection on Day 85.
Period: Overall Study
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Started | 20 | 15 | 5 | 16 | 10
Received Treatment | 19 | 14 | 3 | 15 | 10
Received All Scheduled Treatments | 16 | 13 | 2 | 15 | 10
Completed | 17 | 13 | 2 | 15 | 9
Not Completed | 3 | 2 | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Not Eligible at Randomization | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant: Participants received 0.5 mL cH8/1N1 live-attenuated influenza virus vaccine (LAIV) administered as 0.25 mL drops per nostril on Day 1 followed by 0.5 mL AS03-adjuvanted cH5/1N1 inactivated influenza virus vaccine (IIV) administered as an intramuscular injection on Day 85.
- Total: Total of all reporting groups
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo | Total
Number analyzed (Participants) | 20 | 15 | 5 | 16 | 10 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (5.3) | 27.5 (5.9) | 25.0 (3.7) | 30.3 (5.5) | 29.3 (4.6) | 28.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 2 | 10 | 5 | 41
  Male | 6 | 5 | 3 | 6 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 20 | 13 | 4 | 16 | 10 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 10 | 4 | 14 | 7 | 50
  White | 5 | 3 | 0 | 2 | 3 | 13
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Reactions Within 7 Days Following Each Vaccination
Description: Solicited adverse events were assessed by study staff for 60 minutes after each vaccination and and then by study participants daily for 7 days on a a diary card.
  Solicited local reactions included:
  * Post LAIV dose: nasal congestion, rhinorrhea;
  * Post IIV dose: pain, redness, swelling.
Time Frame: 7 days after each vaccination (Days 1-8 and Days 85-92)
Population: Participants who received the priming dose and booster dose
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
Participants
  Post Prime Dose: Any Local Reacton | 10 | 2 | 0 | 11 | 1
  Post Prime Dose: Nasal Congestion | 4 | 1 | 0 | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection
  Post Prime Dose: Rhinorrhea | 8 | 2 | 0 | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection
  Post Prime Dose: Pain | NA — Reaction not applicable for intranasal administration | NA — Reaction not applicable for intranasal administration | NA — Reaction not applicable for intranasal administration | 11 | 1
  Post Prime Dose: Redness | NA — Reaction not applicable for intranasal administration | NA — Reaction not applicable for intranasal administration | NA — Reaction not applicable for intranasal administration | 1 | 0
  Post Prime Dose: Swelling | NA — Reaction not applicable for intranasal administration | NA — Reaction not applicable for intranasal administration | NA — Reaction not applicable for intranasal administration | 1 | 0
  Post Booster Dose: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Any Local Reacton | 10 | 1 | 0 | 8 | 0
  Post Booster Dose: Nasal Congestion | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection
  Post Booster Dose: Rhinorrhea | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection | NA — Reaction not applicable for intramuscular injection
  Post Booster Dose: Pain | 10 | 1 | 0 | 8 | 0
  Post Booster Dose: Redness | 0 | 0 | 0 | 0 | 0
  Post Booster Dose: Swelling | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited General Reactions Within 7 Days Following Each Vaccination
Description: Solicited adverse events were assessed by study staff for 60 minutes after each vaccination and and then by study participants daily for 7 days on a a diary card.
  Solicited general reactions included:
  * abdominal pain
  * arthralgia
  * cough
  * diarrhea
  * fatigue
  * fever
  * headache
  * myalgia
  * nausea
  * shivering
  * sore throat
  * vomiting
  * wheezing
Time Frame: 7 days after each vaccination (Days 1-8 and Days 85-92)
Population: Participants who received the priming dose and booster dose
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
Participants
  Post Prime Dose: Any General Reaction | 13 | 8 | 1 | 10 | 4
  Post Prime Dose: Fever | 0 | 0 | 0 | 0 | 0
  Post Prime Dose: Shivering | 3 | 0 | 0 | 1 | 0
  Post Prime Dose: Fatigue | 3 | 4 | 0 | 6 | 3
  Post Prime Dose: Headache | 7 | 4 | 1 | 6 | 2
  Post Prime Dose: Myalgia | 4 | 2 | 0 | 6 | 0
  Post Prime Dose: Arthralgia | 0 | 3 | 0 | 2 | 0
  Post Prime Dose: Nausea | 3 | 3 | 0 | 0 | 1
  Post Prime Dose: Vomiting | 1 | 0 | 0 | 0 | 0
  Post Prime Dose: Abdominal Pain | 2 | 2 | 0 | 2 | 2
  Post Prime Dose: Diarrhea | 0 | 0 | 0 | 2 | 1
  Post Prime Dose: Sore Throat | 2 | 1 | 0 | 0 | 0
  Post Prime Dose: Cough | 4 | 0 | 0 | 1 | 0
  Post Prime Dose: Wheezing | 0 | 0 | 0 | 0 | 0
  Post Booster Dose: Any General Reaction: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Any General Reaction | 10 | 5 | 0 | 5 | 1
  Post Booster Dose : Fever: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose : Fever | 0 | 0 | 0 | 0 | 0
  Post Booster Dose: Shivering: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Shivering | 2 | 2 | 0 | 1 | 0
  Post Booster Dose: Fatigue: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Fatigue | 8 | 3 | 0 | 2 | 1
  Post Booster Dose : Headache: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose : Headache | 4 | 4 | 0 | 0 | 1
  Post Booster Dose: Myalgia: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Myalgia | 5 | 1 | 0 | 1 | 0
  Post Booster Dose: Arthralgia: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Arthralgia | 4 | 2 | 0 | 0 | 0
  Post Booster Dose: Nausea: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Nausea | 3 | 2 | 0 | 0 | 0
  Post Booster Dose: Vomiting: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Vomiting | 0 | 0 | 0 | 0 | 0
  Post Booster Dose: Abdominal Pain: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Abdominal Pain | 2 | 1 | 0 | 1 | 0
  Post Booster Dose: Diarrhea: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Diarrhea | 0 | 1 | 0 | 0 | 0
  Post Booster Dose: Sore Throat: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Sore Throat | 3 | 2 | 0 | 0 | 0
  Post Booster Dose: Cough: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Cough | 1 | 1 | 0 | 1 | 0
  Post Booster Dose: Wheezing: number analyzed (Participants) | 16 | 13 | 2 | 15 | 10
  Post Booster Dose: Wheezing | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events Within 28 Days Following Any Vaccination
Description: Unsolicited adverse events (AEs) are any AEs reported spontaneously by the participant, observed by the study personnel during study visits or those identified during review of medical records or source documents, such as diary cards. Participants were asked to record any unsolicited symptoms or other illness description in their diary card during the 28 days after each vaccination.
  All AEs, including clinical laboratory test results, were assessed by a study clinician and the study subject (as applicable) to quantify severity using a protocol-defined grading system as mild (mild symptoms, easily tolerated, not interfering with daily activities), moderate (causing some interference with daily activity), or severe (severe symptoms that prevent normal every day activities).
  The investigator assessed the relationship between study vaccines and the occurrence of each AE using clinical judgment.
Time Frame: 28 days after each vaccination (Days 1 to 28 and Days 85 to 113)
Population: Participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
Participants
  Any adverse events | 10 | 8 | 1 | 6 | 5
  AEs related to study vaccine | 5 | 2 | 0 | 1 | 0
  Mild adverse events | 6 | 3 | 0 | 3 | 3
  Mild AEs related to study vaccine | 5 | 0 | 0 | 0 | 0
  Moderate adverse events | 3 | 4 | 1 | 3 | 2
  Moderate AEs related to study vaccine | 0 | 2 | 0 | 1 | 0
  Severe adverse events | 1 | 1 | 0 | 0 | 0
  Severe AEs related to study vaccine | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Grade 2 or Higher Hematological and Biochemical Laboratory Abnormalities From Day 8 to Day 113
Description: Hematological and biochemical parameters assessed included hemoglobin, platelets, red blood cells, white blood cells (WBC), absolute neutrophil count (ANC), lymphocytes, monocytes, eosinophils, basophils, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, blood urea nitrogen (BUN) and BUN-to-creatinine ratio.
  Grading of laboratory parameters was based on the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials as Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (severe), or Grade 4 (Potentially life-threatening).
  Grade 2 or higher:
  * BUN: > 26 mg/dL
  * Creatinine: > 1.7 mg/dL
  * ALT, AST: > 2.5 × upper limit of normal (ULN)
  * Hemoglobin: < 11.0 g/dL (females) or < 12.5 g/dL (males) or change from baseline > 1.5 g/dL
  * WBC: > 15,000 cell/mm³ or < 2,500 cell/mm³
  * Lymphocytes: < 750 cell/mm³
  * ANC: < 1,500 cell/mm³
  * Eosinophils: > 1,500 cell/mm³
  * Platelets: < 125,000 cell/mm³
Time Frame: Days 8, 29, 85, 92, and 113
Population: Participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
Participants
  Hemoglobin | 0 | 2 | 0 | 3 | 1
  Hemoglobin change from baseline | 3 | 1 | 2 | 3 | 0
  Platelets | 0 | 0 | 0 | 0 | 0
  White blood cell count | 0 | 0 | 0 | 0 | 0
  Absolute neutrophil count | 5 | 1 | 0 | 3 | 0
  Lymphocytes | 0 | 0 | 0 | 0 | 0
  Basophils | 0 | 0 | 0 | 0 | 0
  Monocytes | 0 | 0 | 0 | 0 | 0
  Eosinophils | 1 | 0 | 0 | 0 | 0
  Red blood cells | 0 | 0 | 0 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen | 0 | 0 | 0 | 0 | 0
  BUN to creatinine ratio | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase | 0 | 0 | 0 | 0 | 0
  Asparate aminotransferase | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With a Medically Attended Event (MAE), Laboratory-Confirmed Influenza-like Illness (LC-ILI), Potential Immune-mediated Disease (pIMD), or Serious Adverse Event (SAE) up to Day 113
Description: An MAE is an event for which the participant received medical attention such as hospitalization, an emergency room visit, or a visit to or from medical personnel.
  pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
  LC-ILI is defined as at least 1 systemic symptom (fever or myalgia) AND at least 1 respiratory symptom (cough or sore throat), confirmed by polymerase chain reaction (PCR) assay.
  An SAE is an AE that met any of the following:
  * Death
  * Life threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * Results in congenital anomaly/birth defect
  * An important medical event that may jeopardize the well-being of the subject or require medical or surgical intervention to prevent an above outcome.
Time Frame: Through Day 113 (28 days post-dose 2)
Population: Participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
Participants
  SAEs | 0 | 0 | 1 | 0 | 0
  MAEs | 6 | 2 | 0 | 3 | 1
  LC-ILIs | 0 | 0 | 1 | 0 | 0
  pIMDs | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Any Grade 2 or Higher Hematological and Biochemical Laboratory Abnormalities From Month 9 to Month 15
Description: as for outcome 4
Time Frame: Month 9 (6 months post-dose 2) and Month 15 (12 months post-dose 2)
Population: Participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
Participants
  Hemoglobin | 0 | 1 | 0 | 2 | 0
  Hemoglobin change from baseline | 0 | 1 | 1 | 2 | 0
  Platelets | 0 | 0 | 0 | 0 | 0
  White blood cell count | 1 | 0 | 0 | 0 | 0
  Absolute neutrophil count | 0 | 0 | 0 | 0 | 0
  Lymphocytes | 0 | 0 | 0 | 0 | 0
  Basophils | 0 | 0 | 0 | 0 | 0
  Monocytes | 0 | 0 | 0 | 0 | 0
  Eosinophils | 1 | 0 | 0 | 0 | 0
  Red blood cells | 0 | 0 | 0 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen | 0 | 0 | 0 | 0 | 0
  BUN to creatinine ratio | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase | 0 | 0 | 0 | 0 | 0
  Asparate aminotransferase | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With a Medically Attended Event (MAE), Laboratory-Confirmed Influenza-like Illness (LC-ILI), Potential Immune-mediated Disease (pIMD), or Serious Adverse Event (SAE) up to End of Study
Description: An MAE is an event for which the participant received medical attention such as hospitalization, an emergency room visit, or a visit to or from medical personnel.
  pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
  LC-ILI is defined as at least 1 systemic symptom (fever or myalgia) AND at least 1 respiratory symptom (cough or sore throat), confirmed by PCR assay.
  An SAE is an AE that met any of the following:
  * Death
  * Life threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * Resulted in congenital anomaly/birth defect
  * An important medical event that may jeopardize the well-being of the subject or require medical or surgical intervention to prevent an above outcome.
Time Frame: From first dose to end of study, 588 days (21 months; 18 months post-dose 2)
Population: Participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
Participants
  SAEs | 0 | 0 | 1 | 0 | 2
  MAEs | 7 | 4 | 0 | 4 | 4
  LC-ILIs | 1 | 1 | 1 | 0 | 0
  pIMDs | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants in Groups 1, 2, and 3 With Detectable Influenza A Virus in Nasal and Oropharyngeal Swabs on Days 1 to 5
Description: To detect viral shedding participants who received LAIV vaccine or intranasal sterile saline as the prime dose had nasal and oropharyngeal swabs collected on Days 1 to 5. Influenza type A virus ribonucleic acid (RNA) was detected using reverse transcription polymerase chain reaction (RT-PCR).
Time Frame: Days 1 to 5
Population: Participants who received LAIV (Groups 1, 2, and 3) with evaluable samples
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo
Number analyzed (Participants) | 19 | 14 | 3
Participants
  Overall | 7 | 8 | 0
  Day 2 | 7 | 4 | 0
  Day 3 | 1 | 1 | 0
  Day 4 | 0 | 0 | 0
  Day 5 | 0 | 3 | 0

9. Secondary Outcome: Number of Participants in Groups 1, 2, and 3 With Viable Vaccine Virus in Cell Culture Through 5 Days Post-vaccination
Description: To study virus infectivity, nasal and oropharyngeal swab specimens that tested influenza A positive by RT-PCR were further tested for viability of virus in Madin Darby canine kidney (MDCK) cell culture and stained with monoclonal antibody specific to the cH8/1N1 LAIV virus to confirm detected virus is of vaccine origin.
Time Frame: Days 1 to 5
Population: Participants who received LAIV (Groups 1, 2, and 3) and tested positive for influenza A virus by RT-PCR at any time during the 5 days post LAIV dose and with evaluable samples
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo
Number analyzed (Participants) | 7 | 7 | 0
Participants
  Overall | 0 | 0 |
  Day 2: number analyzed (Participants) | 7 | 3 | 0
  Day 2 | 0 | 0 |
  Day 3: number analyzed (Participants) | 1 | 1 | 0
  Day 3 | 0 | 0 |
  Day 4: number analyzed (Participants) | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 0 | 3 | 0
  Day 5 |  | 0 |

10. Secondary Outcome: Percentage of Participants With Serum Anti-H1 Hemagglutinin Stalk Immunoglobulin G Antibody Seropositivity
Description: Anti-H1 hemagglutinin (HA) stalk immunoglobulin G (IgG) was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]) .
  Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned. Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 65.3 EU/mL.
Time Frame: Baseline (pre-dose 1), Month 1 (28 days post-dose 1), Month 4 (28 days post-dose 2), Month 9 (6 months post-dose 2), and Month 15 (12 months post-dose 2)
Population: Participants in the per-protocol population with available data at each time point. The per protocol population included all participants who received at least 1 vaccination and with no major deviations, including those considered likely to affect the immune response; data were included up to the time of the observed deviation event.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 9 (6 months post-dose 2): number analyzed (Participants) | 15 | 13 | 2 | 14 | 9
  Month 9 (6 months post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

11. Secondary Outcome: Geometric Mean Titer of Serum Anti-H1 Hemagglutinin Stalk IgG Antibodies
Description: Anti-H1 hemagglutinin stalk immunoglobulin G (IgG) was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]) .
  Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned. The lower limit of quantitation (LLOQ) for the assay was 65.3 EU/mL.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
EU/mL
  Baseline (pre-vaccination) | 11503 [7698 to 17187] | 10213 [6559 to 15903] | 12966 [2459 to 68377] | 12028 [6658 to 21729] | 8615 [5517 to 13453]
  Month 1 (28 days post-dose 1) | 11337 [7790 to 16499] | 10347 [6810 to 15721] | 11832 [2593 to 53992] | 84207 [63756 to 111219] | 7975 [5317 to 11961]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 62238 [44507 to 87034] | 22073 [14577 to 33423] | 10628 [NA to 5749922] — < LLOQ (65.3 EU/mL) | 62992 [46931 to 84549] | 9226 [5791 to 14696]
  Month 9 (6 months post-dose 2): number analyzed (Participants) | 15 | 13 | 2 | 14 | 9
  Month 9 (6 months post-dose 2) | 19955 [13334 to 29863] | 10846 [7108 to 16549] | 8364 [NA to 12544501] — < LLOQ (65.3 EU/mL) | 31228 [21153 to 46101] | 7043 [4019 to 12345]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 16046 [10632 to 24218] | 13470 [8300 to 21860] | 16195 | 27323 [17736 to 42092] | 6825 [4132 to 11272]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Adjusted Geometric Mean Titer (GMT) Ratio 28 Days Post-Boost Dose; Test type: Other; p < 0.0001, ANCOVA; GMT Ratio = 2.73, 95% CI 2-sided [1.73 to 4.29] — GMT ratio computed after fitting an analysis of covariance (ANCOVA) model on the log10 transformed titers, including vaccine group as fixed effect and the pre-vaccination titer as covariate
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.9411, ANCOVA; GMT Ratio = 1.06, 95% CI 2-sided [0.68 to 1.66] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p < 0.0001, ANCOVA; GMT Ratio = 0.39, 95% CI 2-sided [0.24 to 0.62] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk IgG Antibodies
Description: Anti-H1 hemagglutinin stalk immunoglobulin G (IgG) was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]) .
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 80.0 [51.9 to 95.7] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 75.0 [47.6 to 92.7] | 15.4 [1.9 to 45.4] | 0.0 [0.0 to 84.2] | 57.1 [28.9 to 82.3] | 0.0 [0.0 to 30.8]
  Month 9 (6 months post-dose 2): number analyzed (Participants) | 15 | 13 | 2 | 14 | 9
  Month 9 (6 months post-dose 2) | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 21.4 [4.7 to 50.8] | 0.0 [0.0 to 33.6]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 7.1 [0.2 to 33.9] | 15.4 [1.9 to 45.4] | 0.0 | 23.1 [5.0 to 53.8] | 0.0 [0.0 to 30.8]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.0025, Fisher Exact; Difference = 59.6, 95% CI 2-sided [23.59 to 81.02]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.4421, Fisher Exact; Difference = 17.9, 95% CI 2-sided [-16.24 to 49.00]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.0461, Fisher Exact; Difference = -41.8, 95% CI 2-sided [-68.75 to -4.80]

13. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk IgG Antibodies
Description: as for outcome 12
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 33.3 [11.8 to 61.6] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 25.0 [7.3 to 52.4] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 30.8]
  Month 9 (6 months post-dose 2): number analyzed (Participants) | 15 | 13 | 2 | 14 | 9
  Month 9 (6 months post-dose 2) | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 33.6]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

14. Secondary Outcome: Mean Geometric Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk IgG Antibodies
Description: Anti-H1 hemagglutinin stalk immunoglobulin G (IgG) was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
  Mean geometric increase represents the fold-rise in antibody titer from baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [0.9 to 1.0] | 1.0 [0.9 to 1.1] | 0.9 [0.8 to 1.1] | 7.0 [4.3 to 11.4] | 0.9 [0.9 to 1.0]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 5.8 [3.8 to 8.8] | 2.2 [1.6 to 3.2] | 1.0 [0.3 to 3.7] | 4.9 [3.2 to 7.5] | 1.1 [0.8 to 1.4]
  Month 9 (6 months post-dose 2): number analyzed (Participants) | 15 | 13 | 2 | 14 | 9
  Month 9 (6 months post-dose 2) | 1.8 [1.4 to 2.3] | 1.1 [0.9 to 1.4] | 0.8 [0.6 to 1.1] | 2.4 [1.7 to 3.5] | 0.8 [0.6 to 1.2]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.5 [1.1 to 1.9] | 1.4 [0.9 to 2.0] | 0.8 | 2.1 [1.5 to 3.0] | 0.8 [0.6 to 1.1]

15. Secondary Outcome: Percentage of Participants With Serum Anti-H1 Hemagglutinin Stalk Immunoglobulin A Antibody Seropositivity
Description: Anti-H1 hemagglutinin stalk immunoglobulin A (IgA) was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgA antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]) .
  Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 1:100.
Time Frame: Baseline (pre-dose 1), Month 1 (28 days post-dose 1), Month 4 (28 days post-dose 2), and Month 15 (12 months post-dose 2)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

16. Secondary Outcome: Geometric Mean Titer of Serum Anti-H1 Hemagglutinin Stalk IgA Antibodies
Description: Anti-H1 hemagglutinin stalk immunoglobulin A (IgA) was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgA antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]) .
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
titer
  Baseline (pre-vaccination) | 5815 [3281 to 10306] | 3536 [1831 to 6826] | 6935 [2425 to 19834] | 3408 [1765 to 6580] | 2887 [1754 to 4753]
  Month 1 (28 days post-dose 1) | 6070 [3585 to 10277] | 4781 [2230 to 10249] | 7824 [1280 to 47812] | 15919 [8635 to 29347] | 3163 [1698 to 5893]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 23595 [15414 to 36116] | 11095 [5304 to 23210] | 7571 [371 to 154530] | 18079 [10319 to 31677] | 2818 [1797 to 4417]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 10267 [5724 to 18417] | 8460 [3625 to 19745] | 5740 | 11856 [5992 to 23458] | 2765 [1546 to 4945]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk IgA (Serum) Humoral Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.1665, ANCOVA; GMT Ratio = 1.71, 95% CI 2-sided [0.84 to 3.48] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgA (Serum) Humoral Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.9377, ANCOVA; GMT Ratio = 1.10, 95% CI 2-sided [0.55 to 2.20] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.3088, ANCOVA; GMT Ratio = 0.64, 95% CI 2-sided [0.31 to 1.33] — [estimate comment as in outcome 11, analysis 1]

17. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk IgA Antibodies
Description: as for outcome 16
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 70.8] | 53.3 [26.6 to 78.7] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 62.5 [35.4 to 84.8] | 46.2 [19.2 to 74.9] | 0.0 [0.0 to 84.2] | 64.3 [35.1 to 87.2] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 14.3 [1.8 to 42.8] | 23.1 [5.0 to 53.8] | 0.0 | 46.2 [19.2 to 74.9] | 0.0 [0.0 to 30.8]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.4667, Fisher Exact; Difference = 16.3, 95% CI 2-sided [-19.85 to 48.88]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p > 0.9999, Fisher Exact; Difference = -1.8, 95% CI 2-sided [-34.76 to 32.17]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Serum) Humoral Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.4495, Fisher Exact; Difference = -18.1, 95% CI 2-sided [-51.15 to 19.37]

18. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk IgA Antibodies
Description: as for outcome 16
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 26.7 [7.8 to 55.1] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 18.8 [4.0 to 45.6] | 15.4 [1.9 to 45.4] | 0.0 [0.0 to 84.2] | 28.6 [8.4 to 58.1] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 30.8]

19. Secondary Outcome: Mean Geometric Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk IgA Antibodies
Description: Anti-H1 hemagglutinin stalk immunoglobulin A (IgA) was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgA antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]) .
  Mean geometric increase represents the fold-rise in antibody titer from baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [0.9 to 1.2] | 1.4 [1.0 to 1.8] | 1.1 [0.5 to 2.7] | 4.7 [2.6 to 8.5] | 1.1 [0.9 to 1.4]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 4.8 [2.9 to 7.9] | 3.4 [2.0 to 5.6] | 0.9 [0.0 to 18.9] | 5.0 [2.8 to 9.1] | 1.0 [0.8 to 1.2]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.8 [1.2 to 2.7] | 2.6 [1.7 to 3.8] | 0.6 | 3.1 [1.6 to 5.9] | 1.0 [0.7 to 1.3]

20. Secondary Outcome: Percentage of Participants With Serum Anti-H1 Hemagglutinin Stalk Neutralizing Antibody Seropositivity
Description: Anti H1 hemagglutinin stalk neutralizing antibodies were quantified using a microneutralization (MN) assay using a virus that expresses a chimeric hemagglutinin that contains an exotic HA head domain (strain A/mallard/Sweden/81/2002 [H6N1]) and the H1 stalk domain (strain A/California/04/2009 [H1N1pandemic]) and an exotic neuraminidase, N5, for which humans are generally naïve (strain: A/mallard/Sweden/86/2003 [H12N5]).
  Seropositivity rate was defined as the percentage of participants with an antibody titer of ≥ 1:10.
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

21. Secondary Outcome: Geometric Mean Titer of Serum Anti-H1 Hemagglutinin Stalk Neutralizing Antibodies
Description: Anti H1 hemagglutinin stalk neutralizing antibodies were quantified using a microneutralization (MN) assay using a virus that expresses a chimeric hemagglutinin that contains an exotic HA head domain (strain A/mallard/Sweden/81/2002 ([H6N1]) and the H1 stalk domain (strain A/California/04/2009 ([H1N1pandemic]) and an exotic neuraminidase, N5, for which humans are generally naïve (strain: A/mallard/Sweden/86/2003 [H12N5]). The LLOQ for the assay was 1:10.
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
titer
  Baseline (pre-vaccination) | 48 [34 to 67] | 49 [29 to 83] | 63 [NA to 881] — < LLOQ (1:10) | 58 [36 to 93] | 43 [25 to 74]
  Month 1 (28 days post-dose 1) | 48 [32 to 72] | 38 [23 to 62] | 50 [NA to 368] — < LLOQ (1:10) | 111 [74 to 166] | 40 [24 to 67]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 153 [103 to 277] | 94 [56 to 157] | 40 [NA to 267306] — < LLOQ (1:10) | 138 [96 to 197] | 37 [24 to 58]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 62 [41 to 96] | 58 [35 to 96] | 80 | 99 [62 to 158] | 40 [25 to 64]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk MN (Serum) Assay: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.0928, ANCOVA; GMT Ratio = 1.61, 95% CI 2-sided [0.94 to 2.77] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk MN (Serum) Assay: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.4198, ANCOVA; GMT Ratio = 1.32, 95% CI 2-sided [0.77 to 2.26] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk MN (Serum) Assay: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.6754, ANCOVA; GMT Ratio = 0.82, 95% CI 2-sided [0.47 to 1.45] — [estimate comment as in outcome 11, analysis 1]

22. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk Neutralizing Antibodies
Description: Anti H1 hemagglutinin stalk neutralizing antibodies were quantified using a microneutralization (MN) assay using a virus that expresses a chimeric hemagglutinin that contains an exotic HA head domain (strain A/mallard/Sweden/81/2002 ([H6N1]) and the H1 stalk domain (strain A/California/04/2009 ([H1N1pandemic]) and an exotic neuraminidase, N5, for which humans are generally naïve (strain: A/mallard/Sweden/86/2003 [H12N5]).
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 5.3 [0.1 to 26.0] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 20.0 [4.3 to 48.1] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 50.0 [24.7 to 75.3] | 30.8 [9.1 to 61.4] | 0.0 [0.0 to 84.2] | 35.7 [12.8 to 64.9] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 7.1 [0.2 to 33.9] | 15.4 [1.9 to 45.4] | 0.0 | 15.4 [1.9 to 45.4] | 0.0 [0.0 to 30.8]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk MN (Serum) Assay: Seroresponse (>4-Fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.4515, Fisher Exact; Difference = 19.2, 95% CI 2-sided [-17.19 to 50.49]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk MN (Serum) Assay: Seroresponse (>4-Fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.4837, Fisher Exact; Difference = 14.3, 95% CI 2-sided [-21.22 to 46.19]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk MN (Serum) Assay: Seroresponse (>4-Fold) Rate 28 Days Post-Boost Dose; Test type: Other; p > 0.9999, Fisher Exact; Difference = -4.9, 95% CI 2-sided [-38.80 to 30.46]

23. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk Neutralizing Antibodies
Description: as for outcome 22
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

24. Secondary Outcome: Mean Geometric Increase From Baseline in Serum Anti-H1 Hemagglutinin Stalk Neutralizing Antibodies
Description: Anti H1 hemagglutinin stalk neutralizing antibodies were quantified using a microneutralization (MN) assay using a virus that expresses a chimeric hemagglutinin that contains an exotic HA head domain (strain A/mallard/Sweden/81/2002 [H6N1]) and the H1 stalk domain (strain A/California/04/2009 [H1N1pandemic]) and an exotic neuraminidase, N5, for which humans are generally naïve (strain: A/mallard/Sweden/86/2003 [H12N5]).
  Mean geometric increase represents the fold-rise in antibody titer from baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [0.8 to 1.3] | 0.8 [0.6 to 1.0] | 0.8 [0.3 to 2.1] | 1.9 [1.5 to 2.5] | 0.9 [0.6 to 1.3]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 3.4 [2.2 to 5.2] | 2.1 [1.4 to 3.1] | 0.7 [0.0 to 57.8] | 2.2 [1.6 to 3.0] | 0.9 [0.7 to 1.1]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.2 [0.9 to 1.6] | 1.3 [0.9 to 1.9] | 0.5 | 1.5 [1.1 to 2.2] | 0.9 [0.6 to 1.4]

25. Secondary Outcome: Serum Antibody-dependent Cell-mediated Cytotoxicity (ADCC) to the H1 Hemagglutinin Stalk
Description: Antibody-dependent cell-mediated cytotoxicity (ADCC) is an immune response leading to lysis of antibody-coated target cells by immune effector cells and is triggered by the interaction between the Fc portion of an antibody and Fc-gamma receptors expressed on immune effector cells.
  This bioluminescent assay measured antibodies to a chimeric hemagglutinin (H6 head domain and H1 stalk domain) virus that mediate ADCC activity via the Fc-receptor. ADCC activity was measured in relative luciferase units (RLU) for serial dilutions of serum samples using a plate reader.
  ADCC activity was expressed by the area under the curve (AUC) of luminescence (RLU) per serial dilution (X-fold serial dilutions).
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: RLU * dilution factor
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
RLU * dilution factor
  Baseline (pre-vaccination): number analyzed (Participants) | 19 | 12 | 3 | 15 | 10
  Baseline (pre-vaccination) | 321389 [91992 to 581362] | 200649 [30810 to 542237] | 486775 [173346 to 566708] | 331849 [227546 to 558058] | 109178 [38622 to 239985]
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 19 | 13 | 3 | 15 | 10
  Month 1 (28 days post-dose 1) | 322530 [70776 to 432268] | 183017 [88548 to 457200] | 693225 [104524 to 807975] | 869805 [606000 to 1327125] | 103919 [32655 to 241028]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 1334738 [875063 to 1801500] | 366815 [188478 to 795829] | 474913 [175000 to 774825] | 863811 [524405 to 1521176] | 65371 [28729 to 307257]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 334076 [132771 to 767038] | 353639 [74637 to 840500] | 708455 [708455 to 708455] | 508248 [368035 to 979896] | 130882 [47973 to 310940]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Serum cH6/1 - ADCC Activity: AUC at 28 Days Post-Boost; Test type: Other; p = 0.0031, Wilcoxon (Mann-Whitney); Difference = 2.93, 95% CI 2-sided [1.56 to 7.49] — Based on log10 AUC, using the Hodges-Lehmann location parameter difference back-transformed to the original scale
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Serum cH6/1 - ADCC Activity: AUC at 28 Days Post-Boost; Test type: Other; p = 0.2048, Wilcoxon (Mann-Whitney); Difference = 1.25, 95% CI 2-sided [0.73 to 2.23] — Based on log10 AUC, using the Hodges-Lehmann location parameter difference back-transformed to the original scale
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Serum cH6/1 - ADCC Activity: AUC at 28 Days Post-Boost; Test type: Other; p = 0.0392, Wilcoxon (Mann-Whitney); Difference = 0.43, 95% CI 2-sided [0.18 to 1.00]

26. Secondary Outcome: Fold-Increase From Baseline in Serum ADCC to the H1 Hemagglutinin Stalk
Description: Antibody-dependent cell-mediated cytotoxicity (ADCC) is an immune response leading to lysis of antibody-coated target cells by immune effector cells and is triggered by the interaction between the Fc portion of an antibody and Fc-gamma receptors expressed on immune effector cells.
  This bioluminescent assay measured antibodies to a chimeric hemagglutinin (H6 head domain and H1 stalk domain) virus that mediate ADCC activity via the Fc-receptor. ADCC activity was measured by the area under the curve (AUC) of luminescence per serial dilution.
Time Frame: as for outcome 15
Population: Participants in the per-protocol population with available data at Baseline and each time point. The-per protocol population included all participants who received at least 1 vaccination and with no major deviations, including those considered likely to affect the immune response; data were included up to the time of the observed deviation event.
Measure: Median (95% Confidence Interval); unit: fold-increase
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 12 | 3 | 15 | 10
fold-increase
  Month 1 (28 days post-dose 1) | 0.9 [0.77 to 1.00] | 1.1 [0.90 to 1.35] | 1.2 [0.60 to 1.66] | 2.4 [1.29 to 4.59] | 1.0 [0.58 to 1.18]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 12 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 3.6 [2.22 to 14.36] | 3.8 [1.33 to 18202.00] | 1.2 [1.01 to 1.37] | 2.3 [1.49 to 4.78] | 1.0 [0.51 to 1.59]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.8 [0.67 to 5.20] | 1.8 [0.79 to 4.27] | 1.25 [1.25 to 1.25] | 1.9 [0.82 to 2.12] | 0.9 [0.76 to 1.69]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Serum cH6/1 - ADCC Activity: Fold Increase in AUC at 28 Days Post-Boost; Test type: Other; p = 0.8243, Wilcoxon (Mann-Whitney); Difference = 1.16, 95% CI 2-sided [0.14 to 4.95] — Based on the Hodges-Lehmann location parameter difference on the log scale then back-transformed to the original scale
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Serum cH6/1 - ADCC Activity: Fold Increase in AUC at 28 Days Post-Boost; Test type: Other; p = 0.2530, Wilcoxon (Mann-Whitney); Difference = 1.74, 95% CI 2-sided [0.67 to 6.06] — Based on the Hodges-Lehmann location parameter difference on the log scale then back-transformed to the original scale
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Serum cH6/1 - ADCC Activity: Fold Increase in AUC at 28 Days Post-Boost; Test type: Other; p = 0.5654, Wilcoxon (Mann-Whitney); Difference = 1.83, 95% CI 2-sided [0.47 to 39.92] — Based on the Hodges-Lehmann location parameter difference on the log scale then back-transformed to the original scale

27. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Serum ADCC to the H1 Hemagglutinin Stalk
Description: as for outcome 26
Time Frame: as for outcome 15
Population: Participants in the per-protocol population with available data at Baseline and each time point. The per-protocol population included all participants who received at least 1 vaccination and with no major deviations, including those considered likely to affect the immune response; data were included up to the time of the observed deviation event.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 12 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 70.8] | 26.7 [7.8 to 55.1] | 10.0 [0.3 to 44.5]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 12 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 50.0 [24.7 to 75.3] | 45.5 [16.7 to 76.6] | 0.0 [0.0 to 84.2] | 42.9 [17.7 to 71.1] | 10.0 [0.3 to 44.5]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 28.6 [8.4 to 58.1] | 27.3 [6.0 to 61.0] | 0.0 | 15.4 [1.9 to 45.4] | 0.0 [0.0 to 30.8]

28. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum ADCC to the H1 Hemagglutinin Stalk
Description: as for outcome 26
Time Frame: as for outcome 15
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 12 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 8.3 [0.2 to 38.5] | 0. [0.0 to 70.8] | 13.3 [1.7 to 40.5] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 12 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 31.3 [11.0 to 58.7] | 45.5 [16.7 to 76.6] | 0.0 [0.0 to 84.2] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 14.3 [1.8 to 42.8] | 18.2 [2.3 to 51.8] | 0.0 | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 30.8]

29. Secondary Outcome: Percentage of Participants With Anti-H1 Hemagglutinin Stalk Salivary IgG Antibody Seropositivity
Description: Anti-H1 hemagglutinin stalk immunoglobulin G (IgG) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies in saliva against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
  Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 1:10.
Time Frame: as for outcome 15
Population: Participants in the per-protocol population with available data at each time point. The per-protocol population included all participants who received at least 1 vaccination and with no major deviations, including those considered likely to affect the immune response; data were included up to the time of the observed deviation event.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 18 | 13 | 3 | 15 | 9
percentage of participants
  Baseline (pre-vaccination) | 94.4 | 84.6 | 66.7 | 86.7 | 88.9
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 18 | 13 | 3 | 15 | 8
  Month 1 (28 days post-dose 1) | 94.4 | 84.6 | 100 | 100 | 87.5
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 9
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 88.9
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 13 | 12 | 1 | 12 | 9
  Month 15 (12 months post-dose 2) | 100 | 91.7 | 100 | 100 | 88.9

30. Secondary Outcome: Geometric Mean Titer of Anti-H1 Hemagglutinin Stalk Salivary IgG Antibodies
Description: Anti-H1 hemagglutinin stalk immunoglobulin G (IgG) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]). The LLOQ for the assay was 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 18 | 13 | 3 | 15 | 9
titer
  Baseline (pre-vaccination) | 40 [24 to 65] | 43 [18 to 103] | 21 [NA to 520] — < LLOQ (1:10) | 55 [24 to 123] | 45 [17 to 121]
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 18 | 13 | 3 | 15 | 8
  Month 1 (28 days post-dose 1) | 31 [21 to 48] | 40 [18 to 91] | 42 [14 to 130] | 155 [67 to 356] | 36 [11 to 114]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 9
  Month 4 (28 days post-dose 2) | 161 [102 to 254] | 131 [49 to 346] | 15 [NA to 1153] — < LLOQ (1:10) | 233 [117 to 462] | 61 [16 to 224]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 13 | 12 | 1 | 12 | 9
  Month 15 (12 months post-dose 2) | 67 [32 to 142] | 51 [22 to 114] | 35 | 168 [76 to 372] | 43 [16 to 119]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk IgG (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.8830, ANCOVA; GMT Ratio = 1.21, 95% CI 2-sided [0.45 to 3.27] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.9238, ANCOVA; GMT Ratio = 0.86, 95% CI 2-sided [0.33 to 2.26] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.6926, ANCOVA; GMT Ratio = 0.71, 95% CI 2-sided [0.26 to 1.97] — [estimate comment as in outcome 11, analysis 1]

31. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Anti-H1 Hemagglutinin Stalk Salivary IgG
Description: Anti-H1 hemagglutinin stalk immunoglobulin G (IgG) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies in saliva against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 18 | 13 | 3 | 15 | 9
percentage of participants
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 18 | 13 | 3 | 15 | 8
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 19.5] | 7.7 [0.2 to 36.0] | 33.3 [0.8 to 90.6] | 40.0 [16.3 to 67.7] | 0.0 [0.0 to 36.9]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 9
  Month 4 (28 days post-dose 2) | 53.3 [26.6 to 78.7] | 41.7 [15.2 to 72.3] | 0.0 [0.0 to 84.2] | 57.1 [28.9 to 82.3] | 12.5 [0.3 to 52.7]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 13 | 12 | 1 | 12 | 9
  Month 15 (12 months post-dose 2) | 23.1 [5.0 to 53.8] | 9.1 [0.2 to 41.3] | 0.0 | 33.3 [9.9 to 65.1] | 0.0 [0.0 to 36.9]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk IgG (Saliva), Mucosal Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.7036, Fisher Exact; Difference = 11.7, 95% CI 2-sided [-25.72 to 45.82]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Saliva), Mucosal Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p > 0.9999, Fisher Exact; Difference = -3.8, 95% CI 2-sided [-37.90 to 31.31]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk IgG (Saliva), Mucosal Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.6951, Fisher Exact; Difference = -15.5, 95% CI 2-sided [-49.56 to 22.79]

32. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Anti-H1 Hemagglutinin Stalk Salivary IgG
Description: as for outcome 31
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 18 | 13 | 3 | 15 | 9
percentage of participants
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 18 | 13 | 3 | 15 | 8
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 19.5] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 70.8] | 13.3 [1.7 to 40.5] | 0.0 [0.0 to 36.9]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 9
  Month 4 (28 days post-dose 2) | 20.0 [4.3 to 48.1] | 16.7 [2.1 to 48.4] | 0.0 [0.0 to 84.2] | 21.4 [4.7 to 50.8] | 12.5 [0.3 to 52.7]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 13 | 12 | 1 | 12 | 9
  Month 15 (12 months post-dose 2) | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 28.5] | 0.0 | 25.0 [5.5 to 57.2] | 0.0 [0.0 to 36.9]

33. Secondary Outcome: Mean Geometric Increase of Anti-H1 Hemagglutinin Stalk Salivary IgG Antibodies
Description: Anti-H1 hemagglutinin stalk immunoglobulin G (IgG) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured IgG antibodies in saliva against the H1 stalk domain by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
  Mean geometric increase represents the fold-rise in antibody titer from baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 18 | 13 | 3 | 15 | 9
fold-rise
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 18 | 13 | 3 | 15 | 8
  Month 1 (28 days post-dose 1) | 0.7 [0.5 to 1.1] | 0.9 [0.5 to 1.7] | 2.0 [0.1 to 51.6] | 2.8 [1.2 to 6.7] | 0.8 [0.4 to 1.4]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 9
  Month 4 (28 days post-dose 2) | 4.0 [2.2 to 7.3] | 3.4 [1.6 to 6.9] | 1.2 [0.0 to 1145.6] | 3.6 [1.5 to 8.4] | 1.6 [0.5 to 5.2]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 13 | 12 | 1 | 12 | 9
  Month 15 (12 months post-dose 2) | 2.0 [1.0 to 4.0] | 1.5 [0.9 to 2.6] | 1.2 | 2.8 [0.9 to 9.1] | 0.8 [0.4 to 1.7]

34. Secondary Outcome: Percentage of Participants With Anti-H1 Hemagglutinin Stalk Secretory IgA Antibody Seropositivity in Saliva
Description: Anti-H1 hemagglutinin stalk secretory immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured secretory IgA antibodies antibodies (actively secreted in the mucosa) against the H1 stalk domain in saliva using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
  Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 1:4.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 19 | 13 | 2 | 14 | 9
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 9 | 9
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 12 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

35. Secondary Outcome: Geometric Mean Titer of Anti-H1 Hemagglutinin Stalk Secretory IgA Antibodies in Saliva
Description: Anti-H1 hemagglutinin stalk secretory immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured secretory IgA antibodies antibodies (actively secreted in the mucosa) against the H1 stalk domain in saliva using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]). The LLOQ for the assay was 1:4.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
titer
  Baseline (pre-vaccination): number analyzed (Participants) | 19 | 14 | 3 | 14 | 8
  Baseline (pre-vaccination) | 86 [52 to 143] | 102 [55 to 190] | 58 [10 to 323] | 221 [148 to 330] | 155 [75 to 332]
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 19 | 13 | 2 | 14 | 9
  Month 1 (28 days post-dose 1) | 80 [48 to 133] | 118 [72 to 193] | 77 [NA to 604449] — < LLOQ (1:4) | 191 [95 to 381] | 119 [46 to 308]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 9
  Month 4 (28 days post-dose 2) | 93 [52 to 166] | 136 [86 to 213] | 47 [NA to 11552] — < LLOQ (1:4) | 201 [116 to 347] | 115 [41 to 324]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 12 | 10
  Month 15 (12 months post-dose 2) | 97 [42 to 224] | 109 [56 to 213] | 87 | 190 [115 to 314] | 105 [37 to 294]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk Secretory IgA (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days post-Boost Dose; Test type: Other; p = 0.3203, ANCOVA; GMT Ratio = 0.65, 95% CI 2-sided [0.32 to 1.33] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk Secretory IgA (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days post-Boost Dose; Test type: Other; p = 0.5009, ANCOVA; GMT Ratio = 0.72, 95% CI 2-sided [0.35 to 1.47] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk Secretory IgA (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days post-Boost Dose; Test type: Other; p = 0.9542, ANCOVA; GMT Ratio = 1.10, 95% CI 2-sided [0.51 to 2.37] — [estimate comment as in outcome 11, analysis 1]

36. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Anti-H1 Hemagglutinin Stalk Secretory IgA Antibodies in Saliva
Description: Anti-H1 hemagglutinin stalk secretory immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured secretory IgA antibodies (actively secreted in the mucosa) against the H1 stalk domain in saliva by using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 14 | 8
percentage of participants
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 19 | 13 | 2 | 14 | 8
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 36.9]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 8
  Month 4 (28 days post-dose 2) | 6.7 [0.2 to 31.9] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 41.0]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 12 | 8
  Month 15 (12 months post-dose 2) | 28.6 [8.4 to 58.1] | 0.0 [0.0 to 26.5] | 0.0 | 0.0 [0.0 to 26.5] | 12.5 [0.3 to 52.7]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk Secretory IgA (Saliva), Mucosal Response: Seroresponse (≥4-fold) Rate 28 Days post-Boost Dose; Test type: Other; p > 0.9999, Fisher Exact; Difference = -1.7, 95% CI 2-sided [-30.62 to 23.79]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; [analysis description as in outcome 36, analysis 1]; Test type: Other; p > 0.9999, Fisher Exact; Difference = 6.7, 95% CI 2-sided [-16.24 to 30.34]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; [analysis description as in outcome 36, analysis 1]; Test type: Other; p = 0.4615, Fisher Exact; Difference = 8.3, 95% CI 2-sided [-19.94 to 36.04]

37. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Anti-H1 Hemagglutinin Stalk Secretory IgA Antibodies in Saliva
Description: as for outcome 36
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 14 | 8
percentage of participants
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 19 | 13 | 2 | 14 | 8
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 36.9]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 8
  Month 4 (28 days post-dose 2) | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 41.0]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 12 | 8
  Month 15 (12 months post-dose 2) | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 26.5] | 0.0 | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 36.9]

38. Secondary Outcome: Mean Geometric Increase From Baseline in Anti-H1 Hemagglutinin Stalk Secretory IgA in Saliva
Description: Anti-H1 hemagglutinin stalk secretory immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured secretory IgA antibodies antibodies (actively secreted in the mucosa) against the H1 stalk domain in saliva using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
  Mean geometric increase represents the fold-rise in antibody titer from Baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 14 | 8
fold-rise
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 19 | 13 | 2 | 14 | 8
  Month 1 (28 days post-dose 1) | 0.9 [0.6 to 1.4] | 1.1 [0.7 to 1.7] | 1.3 [1.1 to 1.6] | 0.8 [0.4 to 1.4] | 0.7 [0.3 to 1.7]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 15 | 12 | 2 | 14 | 8
  Month 4 (28 days post-dose 2) | 0.9 [0.5 to 1.6] | 1.4 [0.9 to 2.3] | 1.1 [0.3 to 5.0] | 0.9 [0.6 to 1.3] | 0.6 [0.3 to 1.2]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 12 | 1 | 12 | 8
  Month 15 (12 months post-dose 2) | 1.1 [0.5 to 2.7] | 1.1 [0.6 to 2.3] | 1.6 | 0.9 [0.7 to 1.3] | 0.7 [0.2 to 2.3]

39. Secondary Outcome: Percentage of Participants With Anti-H1 Hemagglutinin Stalk Total IgA Antibody Seropositivity in Saliva
Description: Anti-H1 hemagglutinin stalk total immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured total IgA antibodies antibodies (secreted through active and passive transfer processes in the mucosa) against the H1 stalk domain in saliva using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
  Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 17 | 14 | 2 | 12 | 9
percentage of participants
  Baseline (pre-vaccination): number analyzed (Participants) | 17 | 14 | 2 | 11 | 7
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 16 | 14 | 2 | 12 | 8
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 13 | 13 | 1 | 12 | 9
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 10 | 13 | 1 | 11 | 9
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

40. Secondary Outcome: Geometric Mean Titer of Anti-H1 Hemagglutinin Stalk Total IgA Antibodies in Saliva
Description: Anti-H1 hemagglutinin stalk total immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured total IgA antibodies antibodies (secreted through active and passive transfer processes in the mucosa) against the H1 stalk domain in saliva using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]). The LLOQ for the assay was 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 17 | 14 | 2 | 12 | 9
titer
  Baseline (pre-vaccination): number analyzed (Participants) | 17 | 14 | 2 | 11 | 7
  Baseline (pre-vaccination) | 364 [175 to 758] | 487 [259 to 916] | 317 [NA to NA] — < LLOQ (1:10), 2.181^12 | 792 [420 to 1494] | 541 [252 to 1162]
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 16 | 14 | 2 | 12 | 8
  Month 1 (28 days post-dose 1) | 369 [198 to 687] | 685 [408 to 1148] | 280 [NA to NA] — < LLOQ (1:10), 3.7115^9 | 849 [477 to 1509] | 321 [81 to 1265]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 13 | 13 | 1 | 12 | 9
  Month 4 (28 days post-dose 2) | 625 [265 to 1477] | 543 [269 to 1094] | 39 | 1149 [662 to 1995] | 672 [204 to 2210]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 10 | 13 | 1 | 11 | 9
  Month 15 (12 months post-dose 2) | 353 [152 to 823] | 527 [330 to 843] | 239 | 966 [507 to 1838] | 401 [116 to 1390]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk Total IgA (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.9164, ANCOVA; GMT Ratio = 1.20, 95% CI 2-sided [0.38 to 3.80] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk Total IgA (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.8642, ANCOVA; GMT Ratio = 0.76, 95% CI 2-sided [0.21 to 2.79] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk Total IgA (Saliva), Mucosal Response: Adjusted GMT Ratio 28 Days Post-Boost Dose; Test type: Other; p = 0.6545, ANCOVA; GMT Ratio = 0.63, 95% CI 2-sided [0.18 to 2.27] — [estimate comment as in outcome 11, analysis 1]

41. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Anti-H1 Hemagglutinin Stalk Total IgA Antibodies in Saliva
Description: Anti-H1 hemagglutinin stalk total immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured total IgA antibodies antibodies (secreted through active and passive transfer processes in the mucosa) against the H1 stalk domain in saliva using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 17 | 14 | 2 | 11 | 7
percentage of participants
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 16 | 14 | 2 | 11 | 7
  Month 1 (28 days post-dose 1) | 12.5 [1.6 to 38.3] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 84.2] | 11.1 [0.3 to 48.2] | 14.3 [0.4 to 57.9]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 13 | 13 | 1 | 11 | 7
  Month 4 (28 days post-dose 2) | 30.8 [9.1 to 61.4] | 23.1 [5.0 to 53.8] | 0.0 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 45.9]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 10 | 13 | 0 | 11 | 7
  Month 15 (12 months post-dose 2) | 30.0 [6.7 to 65.2] | 23.1 [5.0 to 53.8] |  | 0.0 [0.0 to 30.8] | 16.7 [0.4 to 64.1]
Statistical Analysis 1: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 2: cH8/1N1 LAIV and cH5/1N1 IIV; Comparison of Anti-H1 HA-stalk Total IgA (Saliva), Mucosal Response: Seroresponse (>4-Fold) Rate 28 Days Post-Boost Dose; Test type: Other; p > 0.9999, Fisher Exact; Difference = 7.7, 95% CI 2-sided [-27.10 to 40.96]
Statistical Analysis 2: Comparison: Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; Comparison of Anti-H1 HA-stalk Total IgA (Saliva), Mucosal Response: Seroresponse (≥4-fold) Rate 28 Days Post-Boost Dose; Test type: Other; p = 0.1045, Fisher Exact; Difference = 30.8, 95% CI 2-sided [-1.76 to 58.19]
Statistical Analysis 3: Comparison: Group 2: cH8/1N1 LAIV and cH5/1N1 IIV vs Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant; [analysis description as in outcome 41, analysis 2]; Test type: Other; p = 0.2292, Fisher Exact; Difference = 23.1, 95% CI 2-sided [-8.62 to 50.86]

42. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Anti-H1 Hemagglutinin Stalk Total IgA Antibodies in Saliva
Description: as for outcome 41
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 17 | 14 | 2 | 11 | 7
percentage of participants
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 16 | 14 | 2 | 11 | 7
  Month 1 (28 days post-dose 1) | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 41.0]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 13 | 13 | 1 | 11 | 7
  Month 4 (28 days post-dose 2) | 7.7 [0.2 to 36.0] | 7.7 [0.2 to 36.0] | 0.0 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 45.9]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 10 | 13 | 0 | 11 | 7
  Month 15 (12 months post-dose 2) | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 24.7] |  | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 45.9]

43. Secondary Outcome: Mean Geometric Increase From Baseline in Anti-H1 Hemagglutinin Stalk Total IgA Antibodies in Saliva
Description: Anti-H1 hemagglutinin stalk total immunoglobulin A (IgA) in saliva was quantified using an enzyme-linked immunosorbent assay (ELISA).
  The ELISA measured total IgA antibodies (secreted through active and passive transfer processes in the mucosa) against the H1 stalk domain in saliva using a chimeric protein containing an exotic H6 hemagglutinin head domain that the vaccinees have not previously been exposed to (strain A/mallard/Sweden/81/02 [H6N1]) and the same H1 stalk domain as expressed by the vaccine (strain A/California/04/09 [H1N1]).
  Mean geometric increase represents the fold-rise in antibody titer from baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 17 | 14 | 2 | 11 | 7
fold-rise
  Month 1 (28 days post-dose 1): number analyzed (Participants) | 16 | 14 | 2 | 11 | 7
  Month 1 (28 days post-dose 1) | 1.1 [0.6 to 2.2] | 1.4 [0.8 to 2.5] | 0.9 [0.0 to 458.5] | 0.7 [0.4 to 1.4] | 0.6 [0.2 to 2.4]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 13 | 13 | 1 | 11 | 7
  Month 4 (28 days post-dose 2) | 1.7 [0.6 to 4.6] | 1.2 [0.5 to 3.2] | 0.7 | 1.1 [0.7 to 1.8] | 0.9 [0.3 to 2.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 10 | 13 | 0 | 11 | 7
  Month 15 (12 months post-dose 2) | 1.2 [0.3 to 5.0] | 1.2 [0.6 to 2.3] |  | 0.9 [0.5 to 1.6] | 0.8 [0.2 to 2.8]

44. Secondary Outcome: Percentage of Participants With Serum Anti-H2 Full-length Hemagglutinin IgG Antibody Seropositivity
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H2, of which the stalk domain shares about 78% amino acid identity with the H1 vaccine stalk domain.
  Anti-H2 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on A/mallard/Netherlands/5/1999 (H2N9) HA.
  Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned. Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 22.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

45. Secondary Outcome: Geometric Mean Titer of Serum Anti-H2 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H2, of which the stalk domain shares about 78% amino acid identity with the H1 vaccine stalk domain.
  Anti-H2 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on A/mallard/Netherlands/5/1999 (H2N9) HA. Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
EU/mL
  Baseline (pre-vaccination) | 6973 [4596 to 10578] | 6027 [3882 to 9357] | 7354 [4095 to 13206] | 7554 [4005 to 14249] | 5597 [3569 to 8776]
  Month 1 (28 days post-dose 1) | 7079 [4720 to 10616] | 6324 [4106 to 9740] | 6757 [4149 to 11002] | 67191 [50322 to 89715] | 4971 [3179 to 7774]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 39171 [26079 to 58833] | 13584 [8684 to 21250] | 8348 [1232 to 56577] | 41005 [28395 to 59213] | 5493 [3326 to 9072]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 13289 [8311 to 21250] | 10682 [6480 to 17609] | 12289 | 26453 [15699 to 44576] | 6283 [3643 to 10836]

46. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Serum Anti-H2 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H2, of which the stalk domain shares about 78% amino acid identity with the H1 vaccine stalk domain.
  Anti-H2 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on A/mallard/Netherlands/5/1999 (H2N9) HA.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 80.0 [51.9 to 95.7] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 68.8 [41.3 to 89.0] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 84.2] | 71.4 [41.9 to 91.6] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 7.7 [0.2 to 36.0] | 0.0 | 46.2 [19.2 to 74.9] | 0.0 [0.0 to 30.8]

47. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum Anti-H2 Full-length Hemagglutinin IgG Antibodies
Description: as for outcome 46
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 53.3 [26.6 to 78.7] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 25.0 [7.3 to 52.4] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 7.7 [0.2 to 36.0] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

48. Secondary Outcome: Mean Geometric Increase of Serum Anti-H2 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H2, of which the stalk domain shares about 78% amino acid identity with the H1 vaccine stalk domain.
  Anti-H2 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on A/mallard/Netherlands/5/1999 (H2N9) HA.
  Mean geometric increase represents the fold-rise in antibody titer from Baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 0.9 [0.8 to 1.1] | 8.9 [5.2 to 15.1] | 0.9 [0.8 to 1.0]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 5.8 [4.0 to 8.5] | 2.2 [1.7 to 2.9] | 1.1 [0.6 to 1.9] | 5.1 [3.2 to 8.1] | 1.0 [0.8 to 1.2]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 2.0 [1.7 to 2.3] | 1.8 [1.2 to 2.6] | 1.3 | 3.3 [2.2 to 5.0] | 1.1 [0.9 to 1.4]

49. Secondary Outcome: Percentage of Participants With Serum Anti-H9 Full-length Hemagglutinin IgG Antibody Seropositivity
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H9, the stalk domain of which shares about 59% amino acid identity with the H1 vaccine stalk domain.
  Anti-H9 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/chicken/Hong Kong/G9/1997 (H9N2) HA. Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned.
  Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 31.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

50. Secondary Outcome: Geometric Mean Titer of Serum Anti-H9 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H9, the stalk domain of which shares about 59% amino acid identity with the H1 vaccine stalk domain.
  Anti-H9 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/chicken/Hong Kong/G9/1997 (H9N2) HA. Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned. The LLOQ for the assay was 31 EU/mL.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
EU/mL
  Baseline (pre-vaccination) | 10613 [7193 to 15660] | 8703 [5569 to 13603] | 13257 [2295 to 76571] | 10436 [5654 to 19261] | 7981 [5204 to 12240]
  Month 1 (28 days post-dose 1) | 10610 [7246 to 15536] | 8683 [5540 to 13611] | 11641 [2239 to 60530] | 37478 [24971 to 56248] | 7477 [5076 to 11013]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 40587 [26113 to 63083] | 16410 [10647 to 25291] | 11081 [NA to 18410906] — < LLOQ (31 EU/mL) | 41113 [26860 to 62931] | 8244 [5491 to 12377]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 16809 [10261 to 27536] | 12271 [7422 to 20287] | 17996 | 24041 [14625 to 39519] | 7593 [4697 to 12275]

51. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Serum Anti-H9 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H9, the stalk domain of which shares about 59% amino acid identity with the H1 vaccine stalk domain.
  Anti-H9 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/chicken/Hong Kong/G9/1997 (H9N2) HA.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 40.0 [16.3 to 67.7] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 37.5 [15.2 to 64.6] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 84.2] | 50.0 [23.0 to 77.0] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 7.1 [0.2 to 33.9] | 7.7 [0.2 to 36.0] | 0.0 | 23.1 [5.0 to 53.8] | 0.0 [0.0 to 30.8]

52. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum Anti-H9 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H9, the stalk domain of which shares about 59% amino acid identity with the H1 vaccine stalk domain.
  Anti-H9 full-length(ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/chicken/Hong Kong/G9/1997 (H9N2) HA.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

53. Secondary Outcome: Mean Geometric Increase of Serum Anti-H9 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin, subtype H9, the stalk domain of which shares about 59% amino acid identity with the H1 vaccine stalk domain.
  Anti-H9 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/chicken/Hong Kong/G9/1997 (H9N2) HA.
  Mean geometric increase represents the fold-rise in antibody titer from Baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [0.9 to 1.1] | 1.0 [0.9 to 1.1] | 0.9 [0.7 to 1.1] | 3.6 [2.4 to 5.5] | 0.9 [0.9 to 1.0]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 3.8 [2.6 to 5.6] | 1.9 [1.4 to 2.6] | 0.9 [0.2 to 4.0] | 3.7 [2.4 to 5.8] | 1.0 [0.8 to 1.3]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.5 [1.2 to 2.0] | 1.5 [1.0 to 2.1] | 0.7 | 2.2 [1.6 to 3.2] | 1.0 [0.7 to 1.4]

54. Secondary Outcome: Percentage of Participants With Serum Anti-H18 Full-length Hemagglutinin IgG Antibody Seropositivity
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin distantly related to the currently circulating influenza A/H1 viruses, subtype H18, the stalk domain of which shares about 65% amino acid identity with the H1 vaccine stalk domain.
  Anti-H18 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/flat-faced bat/Peru/033/10 (H18N11) HA. Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned.
  Seropositivity rate was defined as the percentage of participants with an antibody titer of at least the cut-off for the assay; ≥ 42.3.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

55. Secondary Outcome: Geometric Mean Titer of Serum Anti-H18 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin distantly related to the currently circulating influenza A/H1 viruses, H18, the stalk domain of which shares about 65% amino acid identity with the H1 vaccine stalk domain.
  Anti-H18 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/flat-faced bat/Peru/033/10 (H18N11) HA. Titers are expressed as ELISA units (EU) per mL and were calculated on the basis of an internal standard to which units were arbitrarily assigned.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
EU/mL
  Baseline (pre-vaccination) | 5764 [3981 to 8345] | 5266 [3463 to 8007] | 6142 [2841 to 13276] | 7585 [3822 to 15052] | 5315 [3444 to 8201]
  Month 1 (28 days post-dose 1) | 6030 [4181 to 8696] | 5463 [3560 to 8384] | 5238 [2788 to 9843] | 30197 [19699 to 46292] | 4977 [3279 to 7553]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 25400 [17546 to 36770] | 9965 [6757 to 14695] | 5178 [297 to 90261] | 30254 [20266 to 45165] | 5702 [3692 to 8807]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 8478 [5693 to 12626] | 6403 [4299 to 9538] | 6783 | 14577 [9190 to 23121] | 4747 [2993 to 7531]

56. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase From Baseline in Serum Anti-H18 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin distantly related to the currently circulating influenza A/H1 viruses, subtype H18, the stalk domain of which shares about 65% amino acid identity with the H1 vaccine stalk domain.
  Anti-H18 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/flat-faced bat/Peru/033/10 (H18N11) HA.
Time Frame: as for outcome 15
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 40.0 [16.3 to 67.7] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 50.0 [24.7 to 75.3] | 15.4 [1.9 to 45.4] | 0.0 [0.0 to 84.2] | 50.0 [23.0 to 77.0] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 7.7 [0.2 to 36.0] | 0.0 | 23.1 [5.0 to 53.8] | 0.0 [0.0 to 30.8]

57. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum Anti-H18 Full-length Hemagglutinin IgG Antibodies
Description: as for outcome 56
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 13.3 [1.7 to 40.5] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 25.0 [7.3 to 52.4] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

58. Secondary Outcome: Mean Geometric Increase of Serum Anti-H18 Full-length Hemagglutinin IgG Antibodies
Description: To determine antibody breadth, assays were performed to measure the induction of cross-reactive IgG antibodies to a Group 1 influenza A virus with a heterosubtypic hemagglutinin distantly related to the currently circulating influenza A/H1 viruses, subtype H18, the stalk domain of which shares about 65% amino acid identity with the H1 vaccine stalk domain.
  Anti-H18 full-length (ecto-domain) hemagglutinin IgG was quantified by ELISA using a recombinant antigen based on Strain A/flat-faced bat/Peru/033/10 (H18N11) HA.
  Mean geometric increase represents the fold-rise in antibody titer from Baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 0.9 [0.7 to 1.1] | 4.0 [2.5 to 6.3] | 0.9 [0.9 to 1.0]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 4.5 [3.1 to 6.7] | 2.0 [1.5 to 2.6] | 0.9 [0.3 to 2.3] | 3.8 [2.4 to 6.0] | 1.1 [0.9 to 1.3]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.4 [1.1 to 1.8] | 1.3 [0.9 to 1.8] | 0.9 | 1.8 [1.2 to 2.8] | 0.9 [0.7 to 1.1]

59. Secondary Outcome: Percentage of Participants With Serum Anti-Human H1N1 Virus Neutralizing Antibody Seropositivity
Description: This assay was performed to measure the neutralizing potential of antibodies against the currently circulating human H1N1 isolate which is similar to the stalk used in study vaccines.
  Anti-human H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Singapore/GP1908/2015 (IVR-180).
  Seropositivity rate was defined as the percentage of participants with an antibody titer of ≥ 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

60. Secondary Outcome: Geometric Mean Titer of Serum Anti-Human H1N1 Virus Neutralizing Antibodies
Description: This assay was performed to measure the neutralizing potential of antibodies against the currently circulating human H1N1 isolate which is similar to the stalk used in study vaccines.
  Anti-human H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Singapore/GP1908/2015 (IVR-180). The LLOQ for the assay was 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
titer
  Baseline (pre-vaccination) | 149 [79 to 279] | 108 [46 to 253] | 63 [NA to 881] — < LLOQ (1:10) | 84 [47 to 148] | 98 [38 to 259]
  Month 1 (28 days post-dose 1) | 172 [89 to 332] | 113 [45 to 285] | 50 [NA to 368] — < LLOQ (1:10) | 175 [98 to 313] | 80 [27 to 233]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 217 [129 to 365] | 129 [56 to 301] | 40 [NA to 267306] — < LLOQ (1:10) | 226 [129 to 396] | 106 [38 to 294]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 113 [54 to 239] | 129 [48 to 347] | 80 | 136 [75 to 247] | 130 [54 to 312]

61. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase in Serum Anti-Human H1N1 Virus Neutralizing Antibodies
Description: This assay was performed to measure the neutralizing potential of antibodies against the currently circulating human H1N1 isolate which is similar to the stalk used in study vaccines.
  Anti-human H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Singapore/GP1908/2015 (IVR-180).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 5.3 [0.1 to 26.0] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 20.0 [4.3 to 48.1] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 25.0 [7.3 to 52.4] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 84.2] | 28.6 [8.4 to 58.1] | 10.0 [0.3 to 44.5]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 7.7 [0.2 to 36.0] | 0.0 | 15.4 [1.9 to 45.4] | 10.0 [0.3 to 44.5]

62. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase From Baseline in Serum Anti-Human H1N1 Virus Neutralizing Antibodies
Description: as for outcome 61
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

63. Secondary Outcome: Mean Geometric Increase of Serum Anti-Human H1N1 Virus Neutralizing Antibodies
Description: This assay was performed to measure the neutralizing potential of antibodies against the currently circulating human H1N1 isolate which is similar to the stalk used in study vaccines.
  Anti-human H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Singapore/GP1908/2015 (IVR-180).
  Mean geometric increase represents the fold-rise in antibody titer from Baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.2 [0.9 to 1.5] | 1.1 [0.9 to 1.3] | 0.8 [0.3 to 2.1] | 2.1 [1.4 to 3.0] | 0.8 [0.6 to 1.1]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 1.8 [1.1 to 2.8] | 1.3 [0.9 to 1.8] | 1.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.4 [1.6 to 3.6] | 1.1 [0.6 to 1.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.0 [0.7 to 1.3] | 1.3 [0.9 to 1.9] | 1.0 | 1.6 [1.0 to 2.5] | 1.3 [0.7 to 2.4]

64. Secondary Outcome: Percentage of Participants With Serum Anti-Avian-Swine H1N1 Virus Neutralizing Antibody Seropositivity
Description: This assay was performed to measure the neutralizing potential of cross-reactive antibodies to a Group 1 influenza against an H1N1 virus isolate that currently circulates in animals and is antigenically different from current human isolates.
  Anti-avian-swine H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Swine/Jiangsu/40/2011 (asH1N1).
  Seropositivity rate was defined as the percentage of participants with an antibody titer of ≥ 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

65. Secondary Outcome: Geometric Mean Titer of Serum Anti-Avian-Swine H1N1 Virus Neutralizing Antibodies
Description: This assay was performed to measure the neutralizing potential of cross-reactive antibodies to a Group 1 influenza against an H1N1 virus isolate that currently circulates in animals and is antigenically different from current human isolates.
  Anti-avian-swine H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Swine/Jiangsu/40/2011 (asH1N1). The LLOQ for the assay was 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
titer
  Baseline (pre-vaccination) | 54 [35 to 83] | 46 [26 to 84] | 63 [NA to 881] — < LLOQ (1:10) | 73 [42 to 128] | 61 [26 to 142]
  Month 1 (28 days post-dose 1) | 56 [34 to 90] | 54 [29 to 100] | 63 [NA to 881] — < LLOQ (1:10) | 127 [79 to 204] | 46 [20 to 106]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 141 [95 to 207] | 72 [40 to 130] | 40 [NA to 267306] — < LLOQ (1:10) | 195 [131 to 290] | 57 [25 to 128]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 69 [42 to 114] | 58 [31 to 109] | 80 | 94 [61 to 143] | 70 [34 to 145]

66. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase in Serum Anti-Avian-Swine H1N1 Virus Neutralizing Antibodies
Description: This assay was performed to measure the neutralizing potential of cross-reactive antibodies to a Group 1 influenza against an H1N1 virus isolate that currently circulates in animals and is antigenically different from current human isolates.
  Anti-avian-swine H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Swine/Jiangsu/40/2011 (asH1N1).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 70.8] | 20.0 [4.3 to 48.1] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 37.5 [15.2 to 64.6] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 84.2] | 28.6 [8.4 to 58.1] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 14.3 [1.8 to 42.8] | 15.4 [1.9 to 45.4] | 0.0 | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 30.8]

67. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase in Serum Anti-Avian-Swine H1N1 Virus Neutralizing Antibodies
Description: as for outcome 66
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

68. Secondary Outcome: Mean Geometric Increase From Baseline in Serum Anti-Avian-Swine H1N1 Virus Neutralizing Antibodies
Description: This assay was performed to measure the neutralizing potential of cross-reactive antibodies to a Group 1 influenza against an H1N1 virus isolate that currently circulates in animals and is antigenically different from current human isolates.
  Anti-avian-swine H1N1 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using Strain A/Swine/Jiangsu/40/2011 (asH1N1).
  Mean geometric increase represents the fold-rise in antibody titer from Baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [0.8 to 1.3] | 1.2 [0.8 to 1.7] | 1.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 1.7 [1.3 to 2.4] | 0.8 [0.6 to 1.0]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 2.8 [1.8 to 4.3] | 1.6 [1.1 to 2.3] | 1.0 [NA to NA] — Confidence interval could not be calculated as the variance was zero | 2.4 [1.7 to 3.5] | 0.9 [0.7 to 1.2]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.4 [1.0 to 2.0] | 1.3 [0.8 to 2.0] | 1.0 | 1.3 [0.9 to 1.8] | 1.1 [0.8 to 1.7]

69. Secondary Outcome: Percentage of Participants With Serum Anti-H5N8 Virus Neutralizing Antibody Seropositivity
Description: This assay was performed to measure the induction of antibodies reactive against the head domain of a group 1 influenza virus with a heterosubtypic hemagglutinin from a recent avian influenza virus. Anti-H5N8 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using a reverse genetics (RG) reassortant virus based on Puerto Rico (PR)/8 for 6 genes with 2 surface proteins: HA and neuraminidase (NA) from A/Gyrfalcon/Washington/41088-6/2014 (H5N8).
  Seropositivity rate was defined as the percentage of participants with an antibody titer of ≥ 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Baseline (pre-vaccination) | 100 | 100 | 100 | 100 | 100
  Month 1 (28 days post-dose 1) | 100 | 100 | 100 | 100 | 100
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 100 | 100 | 100 | 100 | 100
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 100 | 100 | 100 | 100 | 100

70. Secondary Outcome: Geometric Mean Titer of Serum Anti-H5N8 Virus Neutralizing Antibodies
Description: This assay was performed to measure the induction of antibodies reactive against the head domain of a group 1 influenza virus with a heterosubtypic hemagglutinin from a recent avian influenza virus. Anti-H5N8 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using a reverse genetics (RG) reassortant virus based on PR8 for 6 genes with 2 surface proteins: HA and NA from A/Gyrfalcon/Washington/41088-6/2014 (H5N8). The LLOQ for the assay was 1:10.
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
titer
  Baseline (pre-vaccination) | 37 [29 to 48] | 30 [23 to 38] | 40 [NA to 224] — < LLOQ (1:10) | 35 [26 to 47] | 28 [22 to 37]
  Month 1 (28 days post-dose 1) | 36 [27 to 47] | 27 [21 to 35] | 50 [NA to 699] — < LLOQ (1:10) | 55 [40 to 76] | 26 [20 to 34]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 62 [43 to 88] | 47 [37 to 60] | 57 [NA to 30902821] — < LLOQ (1:10) | 66 [49 to 88] | 30 [20 to 46]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 42 [29 to 61] | 34 [25 to 46] | 20 | 55 [38 to 80] | 30 [20 to 46]

71. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase in Serum Anti-H5N8 Virus Neutralizing Antibodies
Description: This assay was performed to measure the induction of antibodies reactive against the head domain of a group 1 influenza virus with a heterosubtypic hemagglutinin from a recent avian influenza virus. Anti-H5N8 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using a reverse genetics (RG) reassortant virus based on PR8 for 6 genes with 2 surface proteins: HA and NA from A/Gyrfalcon/Washington/41088-6/2014 (H5N8).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 12.5 [1.6 to 38.3] | 15.4 [1.9 to 45.4] | 0.0 [0.0 to 84.2] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 15.4 [1.9 to 45.4] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

72. Secondary Outcome: Percentage of Participants With a ≥ 10-fold Increase in Serum Anti-H5N8 Virus Neutralizing Antibodies
Description: as for outcome 71
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
percentage of participants
  Month 1 (28 days post-dose 1) | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 30.8]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 0.0 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 30.8]

73. Secondary Outcome: Mean Geometric Increase From Baseline in Serum Anti-H5N8 Virus Neutralizing Antibodies
Description: This assay was performed to measure the induction of antibodies reactive against the head domain of a group 1 influenza virus with a heterosubtypic hemagglutinin from a recent avian influenza virus. Anti-H5N8 virus neutralizing antibodies were quantified using a microneutralization (MN) assay using a reverse genetics (RG) reassortant virus based on PR8 for 6 genes with 2 surface proteins: HA and NA from A/Gyrfalcon/Washington/41088-6/2014 (H5N8).
  Mean geometric increase represents the fold-rise in antibody titer from Baseline to each post-baseline time point (ratio of post-baseline titer to Baseline titer).
Time Frame: as for outcome 15
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
Number analyzed (Participants) | 19 | 14 | 3 | 15 | 10
fold-rise
  Month 1 (28 days post-dose 1) | 1.0 [0.8 to 1.1] | 0.9 [0.8 to 1.0] | 1.3 [0.5 to 3.4] | 1.6 [1.3 to 2.0] | 0.9 [0.8 to 1.1]
  Month 4 (28 days post-dose 2): number analyzed (Participants) | 16 | 13 | 2 | 14 | 10
  Month 4 (28 days post-dose 2) | 1.8 [1.3 to 2.3] | 1.6 [1.2 to 2.2] | 1.4 [0.0 to 115.6] | 1.9 [1.5 to 2.4] | 1.1 [0.7 to 1.5]
  Month 15 (12 months post-dose 2): number analyzed (Participants) | 14 | 13 | 1 | 13 | 10
  Month 15 (12 months post-dose 2) | 1.1 [0.8 to 1.4] | 1.2 [0.8 to 1.8] | 1.0 | 1.5 [1.2 to 1.9] | 1.1 [0.8 to 1.4]

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were recorded through the end of study, 588 days (21 months). Other adverse events were collected through 28 days after each vaccination (Days 1 to 28 and Days 85 to 113)
Arm/Group | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV | Group 3: Placebo | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant | Group 5: Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/14 | 1/3 | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14 | 1/3 | 0/15 | 2/10
Other Adverse Events (participants affected / at risk) | 10/19 | 8/14 | 1/3 | 6/15 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant (N=19) | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV (N=14) | Group 3: Placebo (N=3) | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant (N=15) | Group 5: Placebo (N=10)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: cH8/1N1 LAIV and cH5/1N1 IIV + Adjuvant (N=19) | Group 2: cH8/1N1 LAIV and cH5/1N1 IIV (N=14) | Group 3: Placebo (N=3) | Group 4: cH8/1N1 IIV + Adjuvant and cH5/1N1 IIV + Adjuvant (N=15) | Group 5: Placebo (N=10)
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Cervicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT03300050/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT03300050/SAP_001.pdf